CLINICAL TRIAL: NCT01508312
Title: Brentuximab Vedotin (SGN-35) in Transplant Eligible Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Seagen Inc. (Industry); Hôpitaux Universitaires Henri Mondor, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-142
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-01

CONDITIONS: Hodgkin's Lymphoma
Keywords: CARBOPLATIN; ETOPOSIDE (VP-16); IFOSFAMIDE; SGN-35 (BRENTUXIMAB VEDOTIN); 11-142
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FDG-PET abnormal (Experimental): Patients will receive 2 cycles of weekly brentuximab vedotin and then undergo evaluation with FDGPET/CT. Patients with normalization of FDG-PET/CT will proceed to ASCT. Patients with persistent abnormalities on FDG-PET/CT will receive 2 cycles of augmented ICE chemotherapy followed by repeat FDG-PET/CT prior to ASCT. Following augmented ICE, patients with negative FDG-PET/CT will proceed to ASCT. Those with persistent abnormalities on FDG-PET/CT will be treated according to their physician's recommendations.
  Interventions: Drug: brentuximab vedotin (SGN-35)
- FDG-PET normalization (Experimental): Patients will receive 2 cycles of weekly brentuximab vedotin and then undergo evaluation with FDGPET/CT. Patients with normalization of FDG-PET/CT will proceed to ASCT. Patients with persistent abnormalities on FDG-PET/CT will receive 2 cycles of augmented ICE chemotherapy followed by repeat FDG-PET/CT prior to ASCT. Following augmented ICE, patients with negative FDG-PET/CT will proceed to ASCT. Those with persistent abnormalities on FDG-PET/CT will be treated according to their physician's recommendations.
  Interventions: Drug: Brentuximab Vedotin (SGN-35)

INTERVENTIONS:
Drug: brentuximab vedotin (SGN-35) — Patients will receive 2 cycles of weekly brentuximab vedotin, 1.2mg/kg on days 1, 8, and 15 of each 28 day cycle. Patients with pre-treatment positive bone marrow biopsies will have repeat bone marrow biopsies if the PET scan is negative. FDG-PET/CT will be repeated after 2 cycles of treatment within 1 week of the last dose of cycle 2. Patients with persistent abnormalities on FDG-PET/CT following 2 cycles of brentuximab vedotin will receive 2 cycles of augmented ICE. The first cycle of augmented ICE will be initiated 7-14 days after the last dose of SGN-35. FDG-PET/CT will be repeated within 7-14 days following the second cycle of augmented ICE. Stem cell mobilization can be performed following the first or second cycle of augmented ICE.
  Arms: FDG-PET abnormal
Drug: Brentuximab Vedotin (SGN-35) — Patients will receive 2 cycles of weekly brentuximab vedotin, 1.2mg/kg on days 1, 8, and 15 of each 28 day cycle. FDG-PET/CT will be repeated after 2 cycles of treatment within 1 week of the last dose of cycle 2. Patients with pre-treatment positive bone marrow biopsies will have repeat bone marrow biopsies if the PET scan is negative. Patients with normalization of FDG-PET/CT and negative bone marrow biopsies following 2 cycles of brentuximab vedotin will undergo stem cell mobilization in preparation for ASCT.
  Arms: FDG-PET normalization

SUMMARY:
The purpose of this study is determine if 2 cycles of SGN-35 can be used instead of ICE prior to autologous stem cell transplant (ASCT) for relapsed and refractory HL. There are 2 steps to treating patients with relapsed or refractory HL. The first step is to shrink the lymphoma with chemotherapy. The chemotherapy regimen commonly used is called ICE. ICE is a combination of chemotherapy drugs: ifosfamide, carboplatin, and etoposide. The second step of treatment is to give high doses of chemotherapy and radiation therapy followed by infusion of stem cells. This is called an ASCT. This study will focus on the first step of treatment for relapsed and refractory HL.

ICE chemotherapy can cause many side effects. We believe that there are patients who can receive less toxic treatments and still do well. We have learned from past studies that [18F]FDG-PET scans (which we will call "PET scans") can be used to predict who will do well after ASCT. PET scans are tests used to measure the metabolic activity of the disease. Patients without abnormal activity on their PET scan (negative PET scan) before ASCT are much more likely to be cured than those with activity on their PET scan (positive PET scan).

In this study, instead of beginning with ICE chemotherapy, the patient will receive a new drug called Brentuximab vedotin (SGN-35). SGN-35 is a type of drug called an antibody drug conjugate. SGN-35 has 2 parts; a part that targets cancer cells (the antibody) and a cell killing part (the chemotherapy). The antibody part of SGN-35 sticks to a target called CD30. CD30 is an important molecule on some cancer cells (including Hodgkin lymphoma) and some normal cells of the immune system. The cell killing part of SGN-35 is a chemotherapy called monomethyl auristatin E (MMAE).

It can kill cells that the antibody part of SGN-35 sticks to.

Compared to ICE chemotherapy, SGN-has fewer side effects and does not require inpatient admission for treatment. We aim to determine whether patients can avoid treatment with ICE prior to ASCT. We will use the results of the PET scan to determine whether the patient needs additional chemotherapy before ASCT. If the PET scan is negative, the patient will be referred to ASCT and not receive ICE chemotherapy. If the PET scan is positive, the physician will discuss further treatment options with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of cd30 positive classical Hodgkin's lymphoma.
* Primary refractory or relapsed disease proven by biopsy or fine needle aspiration (cytology) of an involved site. Pathology must be reviewed at MSKCC.
* Relapse or refractory disease following doxorubicin or nitrogen mustard containing front-line therapy
* Fluorodeoxyglucose (FDG)-avid disease by FDG-PET/CT and measurable disease of at least 1.5 cm by spiral CT, as assessed by the site radiologist.
* Cardiac ejection fraction of greater than 45%, measured since last chemotherapy.
* Hemoglobin-adjusted diffusing capacity for carbon monoxide of greater than 50% on pulmonary function testing, measured since last chemotherapy
* Serum creatinine < or = to 1.5 mg/dl; if creatinine >1.5 mg/dl then the measured 12- or 24-hour creatinine clearance must be >60 ml/minute.
* ANC>1000/μl and Platelets>50,000/μl
* Total bilirubin < 2.0 mg/dl in the absence of a history of Gilbert's disease.
* Females of childbearing age must be on an acceptable form of birth control.
* Age between 12 and 72
* HIV I and II negative.

Exclusion Criteria:

* Received more than 1 prior treatment (combined modality therapy represents 1 treatment) for Hodgkin Lymphoma
* Hepatitis B surface antigen positive or hepatitis B core antibody positive.
* Known pregnancy or breast-feeding.
* Medical illness unrelated to Hodgkin's Lymphoma, which, in the opinion of the attending physician and/or principal investigator, makes participation in this study inappropriate.
* Peripheral neuropathy > grade 2

Ages: 12 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Driessen J, Zwezerijnen GJC, Schoder H, Kersten MJ, Moskowitz AJ, Moskowitz CH, Eertink JJ, Heymans MW, Boellaard R, Zijlstra JM. Prognostic model using 18F-FDG PET radiomics predicts progression-free survival in relapsed/refractory Hodgkin lymphoma. Blood Adv. 2023 Nov 14;7(21):6732-6743. doi: 10.1182/bloodadvances.2023010404. PMID 37722357
- [Derived] Moskowitz AJ, Schoder H, Yahalom J, McCall SJ, Fox SY, Gerecitano J, Grewal R, Hamlin PA, Horwitz S, Kobos R, Kumar A, Matasar M, Noy A, Palomba ML, Perales MA, Portlock CS, Sauter C, Shukla N, Steinherz P, Straus D, Trippett T, Younes A, Zelenetz A, Moskowitz CH. PET-adapted sequential salvage therapy with brentuximab vedotin followed by augmented ifosamide, carboplatin, and etoposide for patients with relapsed and refractory Hodgkin's lymphoma: a non-randomised, open-label, single-centre, phase 2 study. Lancet Oncol. 2015 Mar;16(3):284-92. doi: 10.1016/S1470-2045(15)70013-6. Epub 2015 Feb 13. PMID 25683846
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: FDG-PET Abnormal; Cohort 1: FDG-PET Normalization; Cohort 2, Expansion Cohort: FDG-PET Abnormal; Cohort 2, Expansion Cohort: FDG-PET Normalization: Patients will receive 2 cycles of weekly brentuximab vedotin and then undergo evaluation with FDGPET/CT. Patients with normalization of FDG-PET/CT will proceed to ASCT. Patients with persistent abnormalities on FDG-PET/CT will receive 2 cycles of augmented ICE chemotherapy followed by repeat FDG-PET/CT prior to ASCT. Following augmented ICE, patients with negative FDG-PET/CT will proceed to ASCT. Those with persistent abnormalities on FDG-PET/CT will be treated according to their physician's recommendations.
Period: Overall Study
Arm/Group | Cohort 1: FDG-PET Abnormal | Cohort 1: FDG-PET Normalization | Cohort 2, Expansion Cohort: FDG-PET Abnormal | Cohort 2, Expansion Cohort: FDG-PET Normalization
Started | 33 | 12 | 14 | 6
Completed | 32 | 11 | 10 | 6
Not Completed | 1 | 1 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Participant's Hodgkin's lymphoma relapsed, proven by a biopsy sample. | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: FDG-PET Abnormal | Cohort 1: FDG-PET Normalization | Cohort 2, Expansion Cohort: FDG-PET Abnormal | Cohort 2, Expansion Cohort: FDG-PET Normalization | Total
Number analyzed (Participants) | 33 | 12 | 14 | 6 | 65
Age, Continuous [Mean (Full Range); unit: years] | 31 [17 to 65] | 37 [13 to 64] | 33 [19 to 59] | 39 [28 to 54] | 33 [13 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 9 | 5 | 34
  Male | 17 | 8 | 5 | 1 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 0 | 5
  Not Hispanic or Latino | 30 | 10 | 12 | 6 | 58
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 31 | 9 | 12 | 6 | 58
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 12 | 14 | 6 | 65

OUTCOME MEASURES:

1. Primary Outcome: FDG-PET/CT Standardized Uptake Value at 12 Months
Description: Following salvage therapy with brentuximab vedotin (SGN-35) alone or followed by augmented ICE chemotherapy.
Time Frame: 12 months
Measure: Geometric Mean (95% Confidence Interval); unit: Standardized Uptake Value (SUV)
Arm/Group | Cohort 1: FDG-PET Abnormal | Cohort 1: FDG-PET Normalization | Cohort 2, Expansion Cohort: FDG-PET Abnormal | Cohort 2, Expansion Cohort: FDG-PET Normalization
Number analyzed (Participants) | 33 | 12 | 14 | 6
Standardized Uptake Value (SUV) | 69 [53 to 85] | 27 [13 to 40] | 69 [39 to 91] | 30 [12 to 54]

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate (CR and PR rate) to brentuximab vedotin alone
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: FDG-PET Abnormal | Cohort 1: FDG-PET Normalization | Cohort 2, Expansion Cohort: FDG-PET Abnormal | Cohort 2, Expansion Cohort: FDG-PET Normalization
Number analyzed (Participants) | 33 | 12 | 14 | 6
Participants
  Complete Response/CR | 13 | 0 | 4 | 0
  No CR | 20 | 12 | 10 | 6

3. Secondary Outcome: Participants Evaluated for Toxicity
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: FDG-PET Abnormal | Cohort 1: FDG-PET Normalization | Cohort 2, Expansion Cohort: FDG-PET Abnormal | Cohort 2, Expansion Cohort: FDG-PET Normalization
Number analyzed (Participants) | 33 | 12 | 14 | 6
Participants | 33 | 12 | 14 | 6

ADVERSE EVENTS:
Time Frame: 2 years
Description: Cohort 1: FDG-PET Abnormal and Cohort 2: Expansion Cohort: FDG-PET Abnormal received the same intervention. Cohort 1: FDG-PET Normalization and Cohort 2, Expansion Cohort: FDG-PET Normalization received the same intervention
Arm/Group | FDG-PET Abnormal | FDG-PET Normalization
All-Cause Mortality (participants affected / at risk) | 3/47 | 0/18
Serious Adverse Events (participants affected / at risk) | 21/47 | 3/18
Other Adverse Events (participants affected / at risk) | 47/47 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDG-PET Abnormal (N=47) | FDG-PET Normalization (N=18)
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 3
Infection: Anorectal (Infections and infestations) | 2 | 0
Infection: Skin (Infections and infestations) | 1 | 0
PML/Progressive multifocal leukoencephalopathy (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperglycemia (Investigations) | 0 | 2
Fever (General disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Mental status change (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDG-PET Abnormal (N=47) | FDG-PET Normalization (N=18)
Fatigue (General disorders) | 30 | 14
Hyperglycemia (Investigations) | 31 | 12
AST increase (Investigations) | 28 | 12
ALT increase (Investigations) | 27 | 13
Rash (Skin and subcutaneous tissue disorders) | 26 | 14
Neuropathy (Nervous system disorders) | 22 | 6
Alk Phos increased (Investigations) | 18 | 4
Constipation (Gastrointestinal disorders) | 14 | 7
White blood cell decreased (Investigations) | 14 | 5
Nausea (Gastrointestinal disorders) | 13 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 10 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 3
Platelet count decreased (Investigations) | 8 | 5
Hypernatremia (Metabolism and nutrition disorders) | 7 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Neutrophil count decreased (Investigations) | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 3
Lymphocyte count decreased (Investigations) | 5 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT01508312/Prot_SAP_000.pdf